CLINICAL TRIAL: NCT02958722
Title: CO2 or Physiological Solution as Distension Medium: Which One is Better in Diagnostic Hysteroscopy?
Brief Title: Comparison Between Two Different Distention Medium in Diagnostic Hysteroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: ISC2
Record Dates: First submitted 2016-10-21; First posted 2016-11-08 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2016-11

CONDITIONS: Hysteroscopy, Distension Medium, Pain
MeSH Terms: conditions — Pain | interventions — Hysteroscopy; Carbon Dioxide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- carbon dioxide (Active Comparator): Diagnostic hysteroscopy performed with the carbon dioxide (gas)
  Interventions: Procedure: diagnostic hysteroscopy; Drug: carbon dioxide
- physiological solution (Active Comparator): Diagnostic hysteroscopy performed with liquid solution (physiologic solution)
  Interventions: Procedure: diagnostic hysteroscopy; Drug: physiological solution

INTERVENTIONS:
Procedure: diagnostic hysteroscopy — Endoscopic procedure to visualize uterine cavity
Drug: physiological solution
  Arms: physiological solution
Drug: carbon dioxide
  Arms: carbon dioxide

SUMMARY:
The investigators aim to enroll 2000 patients to undergo diagnostic hysteroscopy for suspected uterine pathologies. Women will be randomized into two groups on the basis of distension medium : group A CO2; group B physiological solution. Pain discomfort will be evaluated after the examination.

ELIGIBILITY:
Inclusion Criteria:

* suspected uterine pathologies
* infertility

Exclusion Criteria:

* pregnancy
* severe hypertension, cardiovascular disease or respiratory disease

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Actual)
Dates: Start 2016-11; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
pain discomfort during the procedure assessed through visual analogue scale (VAS) | up to six months

IPD SHARING:
Plan to Share IPD: No